CLINICAL TRIAL: NCT03527563
Title: A Comparative Study on Internet Medical Models and Conventional Medical Models for the Management of Patients With Hypertension in China
Brief Title: Study on Internet Medical Models for the Management of Patients With Hypertension in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Cardiovascular Association (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The study is a multi-center, randomized, open, and parallel study. Approximately 958 subjects will be enrolled in 16 sites. The random number table will be adopted to conduct cluster randomization per township hospital/community health service center. Patients will be randomized 1:1 to receive blood pressure management in Internet medical model or Conventional medical model. After follow-ups of 3 months and 6 months, the blood pressure in each group will be observed and compared
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet Medical Model (Other): Using Internet blood pressure management model: home blood pressure self-monitoring + Internet diagnosis + Maintained or adjusted anti-hypertension drug(s) treatment.
  Interventions: Behavioral: Internet Medical Model
- Conventional Medical Model (No Intervention): Using Conventional blood pressure management model: home blood pressure monitoring + face-to-face diagnosis in clinic + Maintained or adjusted anti-hypertension drug(s) treatment.

INTERVENTIONS:
Behavioral: Internet Medical Model — Subjects in the Internet group should upload blood pressure monitoring data at least once per day. It is highly recommended to upload two pressure monitoring results to capture more blood pressure information. The warning value of blood pressure set in the cloud database is systolic blood pressure ≥ 180mmHg or ≤ 100mmHg and diastolic blood pressure ≥ 110mmHg or ≤ 60mmHg. After enrollment, subjects and physicians communicate via telephone or Internet every two weeks until blood pressure is well controlled judged by physician. Then the frequency of communication will be changed to once a month. Once there are lacks of blood pressure data in 3 days of each week, or. blood pressure values of the subject exceed the warning value in 2 days of consecutive 3 days, the physician will take the initiative to contact the patient for disease inquiry.
  Arms: Internet Medical Model

SUMMARY:
The study is a multi-center, randomized, open, and parallel study. Approximately 958 subjects will be enrolled in 16 sites. The random number table will be adopted to conduct cluster randomization per township hospital/community health service center. Patients will be randomized 1:1 to receive blood pressure management in Internet medical model or Conventional medical model. After follow-ups of 3 months and 6 months, the blood pressure in each group will be observed and compared.

DETAILED DESCRIPTION:
Protocol Title：A Comparative Study on Internet Medical Models and Conventional Medical Models for the Management of Patients with Hypertension in China Study Indication:Hypertension Number of Site:16sites Study Duration (from the initiation of the first site to the end of the follow-up for the last subject): 12 months Duration of Treatment and Management: 6 months Planned Number of Subjects:958 subjects, 479 in each group(blood pressure management in Internet medical model, Conventional medical model) Internet Medical Model:Using Internet blood pressure management model: home blood pressure self-monitoring + Internet diagnosis + Maintained or adjusted anti-hypertension drug(s) treatment.

Conventional Medical Model:Using Conventional blood pressure management model: home blood pressure monitoring + face-to-face diagnosis in clinic + Maintained or adjusted anti-hypertension drug(s) treatment.

Inclusion Criteria：

1. Male or female, 45 to 75 years old (including 45and 75 years);
2. Two measurements of resting systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg on different days during screening;
3. Female subjects of child-bearing potential who are willing to adopt one of the following methods for contraception during the study:

   * Oral contraceptive, either combined or progestogen alone.
   * Injectable progestogen.
   * Implants of levonorgestrel.
   * Oestrogenic vaginal ring.
   * Percutaneous contraceptive patches.
   * Intrauterine device or intrauterine system showing that the expected failure rate is less than 1% per year as stated in the product label.
   * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).
4. Subjects who can understand and perform home blood pressure monitoring as required by the study;
5. Subjects who voluntarily participate in the study and sign informed consent form.

Exclusion Criteria：

1. Two measurements of resting systolic blood pressure ≥ 180mmHg and/or diastolic blood pressure ≥ 110mmHg on different days during screening;
2. Subjects with the history of cerebral stroke within 6 months prior to screening;
3. Subjects with the history of myocardial infarction within 6 months prior to screening;
4. Subjects with the history of heart failure;
5. Subjects with the history of atrial fibrillation;
6. Subjects with the history of coronary artery revascularization;
7. Subjects with other serious diseases, such as tumor;
8. Subjects diagnosed as the secondary hypertension;
9. Subjects with congenital or acquired organic heart disease;
10. Pregnant or lactant subjects;
11. Subjects with severe mental disease;
12. Subjects with abnormal liver and renal function: ALT or AST>2 X upper limit value; Or creatinine > 2X upper limit value
13. Subjects who were previously diagnosed with diabetes that is currently poorly controlled: FBG>10mmol/L;
14. Subjects who are unable to conduct blood pressure self-test;
15. The subject has any other known condition at screening that would compromise subject safety, might affect life expectancy, or making it difficult to successfully manage and follow the subject according to the protocol.

Efficacy Evaluations：

Primary Efficacy Endpoints:

* Blood pressure control rate of subjects in the two groups at Month 6 Secondary Efficacy Endpoints：
* Blood pressure control rate of subjects in the two groups at Month 3
* Blood pressure value of subjects in the two groups at Month 3 and Month 6
* Change of blood pressure of subjects in the two groups at Month 3 and Month 6
* Variability of blood pressure of subjects in the two groups at Month 3 and Month 6
* Treatment compliance of subjects in the two groups at Month 3 and Month 6
* Medical expense of subjects in the two groups at Month 3 and Month 6
* Treatment satisfaction of subjects in the two groups at Month 3 and Month 6

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 45 to 75 years old (including 45 and 75 years);
2. Two measurements of resting systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg on different days during screening;
3. Female subjects of child-bearing potential who are willing to adopt one of the following methods for contraception during the study:

   Oral contraceptive, either combined or progestogen alone. Injectable progestogen. Implants of levonorgestrel. Oestrogenic vaginal ring. Percutaneous contraceptive patches. Intrauterine device or intrauterine system showing that the expected failure rate is less than 1% per year as stated in the product label.

   Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).
4. Subjects who can understand and perform home blood pressure monitoring as required by the study;
5. Subjects who voluntarily participate in the study and sign informed consent form.

Exclusion Criteria:

1. Two measurements of resting systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥110mmHg on different days during screening;
2. Subjects with the history of cerebral stroke within 6 months prior to screening;
3. Subjects with the history of myocardial infarction within 6 months prior to screening;
4. Subjects with the history of heart failure;
5. Subjects with the history of atrial fibrillation;
6. Subjects with the history of coronary artery revascularization;
7. Subjects with other serious diseases, such as tumor;
8. Subjects diagnosed as the secondary hypertension;
9. Subjects with congenital or acquired organic heart disease;
10. Pregnant or lactant subjects;
11. Subjects with severe mental disease;
12. Subjects with abnormal liver and renal function: ALT or AST>2 X upper limit value; Or creatinine >2 X upper limit value;
13. Subjects who were previously diagnosed with diabetes that is currently poorly controlled: FBG>10mmol/L;
14. Subjects who are unable to conduct blood pressure self-test;
15. The subject has any other known condition at screening that would compromise subject safety, might affect life expectancy, or making it difficult to successfully manage and follow the subject according to the protocol.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 958 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: blood pressure control rate of subjects in the two groups at Month 6 | 6 months
  Definition of blood pressure control rate is that the percent of subjects with systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg

CONTACTS AND LOCATIONS:
Overall Officials: huo yong, master, Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pickering TG, Miller NH, Ogedegbe G, Krakoff LR, Artinian NT, Goff D; American Heart Association; American Society of Hypertension; Preventive Cardiovascular Nurses Association. Call to action on use and reimbursement for home blood pressure monitoring: a joint scientific statement from the American Heart Association, American Society of Hypertension, and Preventive Cardiovascular Nurses Association. J Cardiovasc Nurs. 2008 Jul-Aug;23(4):299-323. doi: 10.1097/01.JCN.0000317429.98844.04. PMID 18596492
- [Result] Lawes CM, Vander Hoorn S, Rodgers A; International Society of Hypertension. Global burden of blood-pressure-related disease, 2001. Lancet. 2008 May 3;371(9623):1513-8. doi: 10.1016/S0140-6736(08)60655-8. PMID 18456100